CLINICAL TRIAL: NCT06861452
Title: RR001 in Combination With Chemotherapy for Patients With Locally Advanced Pancreatic Adenocarcinoma: Open-label, Non-randomized Dose Escalation Phase I/IIa Study
Brief Title: Phase I/IIa Study: RR001 Administered Following Chemotherapy Cycles for Patients With Locally Advanced Pancreatic Carcinoma
Acronym: SNIPER
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: EIR Biotherapies s.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SNIPER; 2024-516019-26-00 (EU CTIS Number)
Record Dates: First submitted 2025-01-28; First posted 2025-03-06 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Locally Advanced Pancreatic Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RR001 Dose Level 1 (Experimental): Treatment consists of two cycles of Nab-PTX 125 mg/mq followed by GEM 1000 mg/mq administered on days 1, 8, and 15, every 28 days. At the end of the 2 cycles patients will undergo to an intra-tumoral administration of RR001 at Dose Level (DL) 1: 80 x 10^6 cells
  Interventions: Drug: RR001
- RR001 Dose Level 2 (Experimental): Treatment consists of two cycles of Nab-PTX 125 mg/mq followed by GEM 1000 mg/mq administered on days 1, 8, and 15, every 28 days. At the end of the 2 cycles patients will undergo to an intra-tumoral administration of RR001 at Dose Level (DL) 2: 160 x 10^6 cells
  Interventions: Drug: RR001
- RR001 Dose Level 3 (Experimental): Treatment consists of two cycles of Nab-PTX 125 mg/mq followed by GEM 1000 mg/mq administered on days 1, 8, and 15, every 28 days. At the end of the 2 cycles patients will undergo to an intra-tumoral administration of RR001 at Dose Level (DL) 3: 240 x 10^6 cells
  Interventions: Drug: RR001

INTERVENTIONS:
Drug: RR001 — RR001, a cell-based gene therapy administered following administration of chemotherapy (Nab-PTX 125 mg/mq and GEM 1000 mg/mq)

SUMMARY:
RR001, a cell-based gene therapy administered following chemotherapy cycles for the treatment of patients with locally advanced pancreatic cancer. Phase I /IIa clinical trial (open label and non-randomized) to test the effects (safety & efficacy) of increasing doses of RR001

DETAILED DESCRIPTION:
This study is intended for people diagnosed with locally advanced pancreatic ductal adenocarcinoma.

Currently, surgical resection is the only treatment that offers a chance to cure this type of tumor, but only a few percentage of locally advanced pancreatic adenocarcinoma patients is able to benefit from this approach. Thus, research is aimed at identifying new treatment strategies based on innovative approaches that can increase the number of people who can access surgery as radically as possible.

The SNIPER study aims to evaluate for the first time in humans the applicability and safety of a new drug (called RR001) based on autologous cells, that are, cells taken from the same subject who receives them. These cells are derived from adipose tissue and are genetically modified to deliver a potent anti-cancer death ligand normally produced by the body with the role to kill tumoral cells.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed pancreatic ductal adenocarcinoma classified as locally advanced pancreatic adenocarcinoma (LPAC)
* Patients with no evidence of peritoneal or hematogenous metastasis
* Patients classified as non-resectable locally advanced pancreatic carcinoma (LAPC) based on imaging (TC and NMR), on multidisciplinary staff evaluation by at least an oncologist, radiologist and a qualified digestive surgeon and accounting for AJCC/UICC TNM and clinical staging
* Measurable tumor according RECIST criteria v 1.1
* Low tumor burden with at least one lesion equal/less than 3,5 cm that is suitable for US guided injection (and needle biopsy).
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2
* Patients must be eligible for chemotherapy treatment (based on standard of care)
* Patient older than 18 years of age
* Adequate hepatic and kidney function/Safe hematologic profile
* Negative serum pregnancy test for females of childbearing potential within days of starting treatment
* Willingness and ability to comply with the scheduled visits, treatment plan, imaging procedures, laboratory tests and other study procedures, including lipoaspirate collection (liposuction)

Exclusion Criteria:

* Patient with pancreatic cystic tumor or pancreatic pseudocyst
* Patient with pancreatic tumor different from adenocarcinoma (endocrine, metastases)
* Patients with unknown stage or recurrent pancreatic cancer
* Patients with immunosuppression or susceptibility to viral infection
* Patients with HIV, hepatitis B, hepatitis C, HTLV-I/II, Treponema Pallidum infections
* Patients with liver cirrhosis or other documented liver diseases
* Patient contraindication to use chemotherapy treatments
* Previous of radiotherapy and chemotherapy for PDAC
* Previous hematopoietic stem cell or organ transplantation
* Irreversible cardiac arrhythmias requiring permanent medication
* Heart insufficiency (> grade II, New York Heart Association NYHA criteria)
* History within the last year of acute or subacute coronary syndromes including myocardial infarction, unstable or severe stable angina pectoris
* Uncontrolled hypertension
* Other malignancies within the past 2 years (not including basal cell carcinoma of the skin, prostate cancer or in situ cervix carcinoma, in situ melanoma).
* Active autoimmune disease
* Use of any investigational agents within 21 days from the administration of study treatment
* Patient has had major open surgery prior to the administration of study treatment
* Uncontrolled intercurrent illness including but not limited to psychiatric illness/social situations that in the opinion of the Investigator would compromise compliance of study requirements or put the patient at unacceptable risk
* Suspected or known allergy or hypersensitivity to fluoroquinolones including but not limited to ciprofloxacin
* Suspected or known allergy or hypersensitivity to protamine sulfate or protamine containing products. Including but not limited to patients who have previously undergone procedures such as coronary angioplasty or cardio-pulmonary bypass, which may involve the use of protamine, diabetics who have been treated with protamine insulin, patients allergic to fish, and men who have undergone a vasectomy or are infertile and may have antibodies to protamine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2026-07-29 (Estimated); Study Completion 2027-01-29 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Safety in terms of monitoring of systemic tolerance, Adverse Events (AEs) and severe AEs (SAEs) assess by CTCAE (Version 5.0) | From the signing of the informed consent onwards and during every visit till the End of Study (EOS) (90±7 days after RR001 delivery) for a total of 26 weeks

SECONDARY OUTCOMES:
Evaluation of feasibility through the assessment of the production capacity of the Cell Factory participating in the study of an adequate quantity of autologous cellular product lots sufficient to treat 80% of the patients recruited | From Day 1 till RR001 delivery (46-57 days)
Evaluation of the Efficacy of the Drug Product: Overall response rates (ORR) | 21 days post RR001 delivery
  Overall response rates (ORR) per RECIST 1.1 criteria till End Of Treatment (EOT)
Evaluation of the Efficacy of the Drug Product: percentage of pathological resection | At Day 24 post RR001 delivery
  Percentage of patient undergoing surgery and percentage of pathological resection
Evaluation of the Efficacy of the Drug Product : Time to progression (TTP) till end of study | Day 90± 7 days post RR001 delivery
Evaluation of the Efficacy of the Drug Product : Progression free survival (PFS) till end of study | Day 90± 7 days post RR001 delivery
Evaluation of the Efficacy of the Drug Product : Overall survival (OS) till end of study | Day 90± 7 days post RR001 delivery
Evaluation of the Efficacy of the Drug Product : Tumoral markers evaluation | Day 90±7 days post RR001 delivery
  Tumoral markers evaluation CA 19.9, CEA till end of study
Evaluation of the Efficacy of the Drug Product : Quality of Life (QoL) Questionnaire of European Organization for Research and Treatment of Cancer (EORTC) - EORTC QLQ-C30 | Day 90± 7 days post RR001 delivery
  Questionnaire on Quality of Life (QoL) collected till the end of the study. The EORTC Quality of Life Group (QLG) Core Questionnaire (EORTC QLQ-C30) is a 30 item instrument meant to assess some of the different aspects that define the QoL of cancer patients.
  The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items.
  Each of the multi-item scales includes a different set of items - no item occurs in more than one scale.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
  Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Evaluation of the Efficacy of the Drug Product : Quality of Life (QoL) Questionnaire of European Organization for Research and Treatment of Cancer (EORTC) - EORTC QLQ-PAN26 | Day 90± 7 days post RR001 delivery
  Questionnaire on Quality of Life collected till the end of the study EORTC QLQ-PAN26 (Pancreatic Cancer Module).
  This questionnaire is administered on the same module of EORTC QLQ-C30 Questionnaire.
  The module comprises 26 questions assessing pain, dietary changes, jaundice, altered bowel habit, emotional problems related to pancreatic cancer, and other symptoms (cachexia, indigestion, flatulence, dry mouth, taste changes).
  All of the scales and single-item measures range in score from 0 to 100, where zero corresponds to the lowest possible score and 100 to the highest possible score.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero-Universitaria (AOU) Policlinico di Modena, Modena, Italy, Italy

IPD SHARING:
Plan to Share IPD: Undecided